CLINICAL TRIAL: NCT02394132
Title: A Randomised Controlled Multicentre Trial of Imiquimod Versus Radiotherapy for Lentigo Maligna (LM) When Staged Surgical Excision With 5mm Margins is Not Possible, is Refused, or Fails
Brief Title: Radiotherapy or Imiquimod in Complex Lentigo Maligna
Acronym: RADICAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02.12
Record Dates: First submitted 2015-03-10; First posted 2015-03-20 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Lentigo Maligna
Keywords: Lentigo maligna; Imiquimod; Radiotherapy
MeSH Terms: conditions — Hutchinson's Melanotic Freckle | interventions — Imiquimod; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imiquimod (Experimental): Topical imiquimod 5% cream
  * application to treatment area for 5 days/week for a total of 12 weeks
  * dispensed at baseline visit along with patient diary
  Interventions: Drug: Imiquimod
- Radiotherapy (Experimental): Radiotherapy
  * treatment regimen determined by treating radiation oncologist and as per standard practice at local institution
  * treatment to commence within 8 weeks of randomisation
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Imiquimod
  Other Names: Aldara
  Arms: Imiquimod
Radiation: Radiotherapy
  Arms: Radiotherapy

SUMMARY:
The purpose of this study is to investigate the effectiveness of using either radiotherapy (RT) or Imiquimod (ImiQ) to treat the Lentigo Maligna (LM), when surgery is not possible, is refused, or fails.

DETAILED DESCRIPTION:
Surgery is the standard treatment for people diagnosed with LM. However for some people, it may not be possible due to the location of their LM lesion(s).

Currently, the Australian and New Zealand Melanoma Treatment Guidelines recommend radiotherapy for the treatment of LM however there is no clinical trial evidence for this and a trial is needed to prove which treatment is safer and more effective. Some clinicians may also recommend the use of a cream called Imiquimod. It is approved and widely used in Australia to treat solar keratosis, superficial basal cell carcinoma, external genital warts, and perianal warts. Although not currently licensed for treatment use in LM, there is some evidence to suggest that it is both safe and effective in treating LM.

This trial will scientifically evaluate and compare these two treatments in a controlled clinical setting.

The primary objective of this trial is to compare the rate of LM treatment failure and recurrence rate measured at 24 months (primary endpoint), and measured at 6, 12 months (secondary endpoints) following treatment with ImiQ or RT. For this study, treatment failure includes both the recurrence and persistence of LM, and is defined as the presence of LM cells within the original field of treatment confirmed by histopathology.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. A biopsy-proven LM. This includes previous treatment failures (not with imiquimod or RT) of LM that are diagnosed as biopsy-proven LM.
3. LM that is in a location amenable to treatment with imiquimod and radiotherapy.
4. Willing and able to comply with study requirements.
5. Written informed consent.

Exclusion Criteria:

1. Invasive melanoma.
2. Medical or psychiatric condition that compromises the ability of the patient to complete protocol treatment or follow-up assessments.
3. Patients who are pregnant or lactating. Women of child bearing potential must have a confirmed negative urine pregnancy test at study entry.
4. Life expectancy of less than 2 years.
5. Radiotherapy sensitivity syndrome

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing LM treatment failure | 6 months
  Determined by systematic biopsy, 6 months following completion of treatment.

SECONDARY OUTCOMES:
LM treatment failure at 12 months and 24 months after the completion of treatment. | 12 and 24 months
  Determined by dermoscopy and/or Reflectance Confocal Microscopy and confirmed by biopsy
Quality of life using Skindex-16 questionnaire | 0-24 months
  Patient Reported outcomes were collected using the dermatology specific quality of life instrument Skindex-16 with additional questions specifically selected from the Skindex-29.
  The Skindex-16 instrument covers three domains: Symptoms, 4 items; Function, 5 items; Emotions, 7 items. Standard scoring of domain scores uses the average of the component items, transformed to 0-100 scale, with higher scores indicating a greater negative impact of skin disease on quality of life (function, emotions) and greater symptom experience.
Quality of life using Skindex-29 questionnaire | 0-24 months
  Due to the nature of this study it was decided to include additional questions from the Skindex-29 instrument (Q2, Q9 and Q18) as these questions address potential issues not covered by the Skindex-16.Similar to the Skindex-16, all responses are transformed to a linear scale of 100, with higher scores indicating more negative impact.
Cosmetic outcome 24 months after treatment or at treatment failure | 24 months
  Evaluated using photographs taken of LM lesion(s) during the study
Incidence of invasive melanoma within treatment fields; a sub-study to evaluate the utility of reflectance confocal microscopy (RCM) compared with standard biopsy in diagnosing recurrence | 0-24 months
  Assessed at all time-points (6, 12 and 24 months post treatment). Time to failure of LM treatment and diagnosis with invasive melanoma within the treatment field was compared for each treatment arm using the log-rank test and Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Guitera, Principal Investigator — Melanoma Institute Australia
Locations (10):
- Australia (8):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Skin and Cancer Foundation, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - St Vincent's Hospital, Sydney, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Hospital das Clinicas, University of Sao Paulo, São Paulo, Brazil
- North Shore Hospital, Takapuna, Auckland, New Zealand